CLINICAL TRIAL: NCT01101035
Title: A Multicenter, Randomized, Active-Control, Phase 3B Study to Evaluate the Cardiovascular Safety of Febuxostat and Allopurinol in Subjects With Gout and Cardiovascular Comorbidities
Brief Title: Cardiovascular Safety of Febuxostat and Allopurinol in Participants With Gout and Cardiovascular Comorbidities (CARES)
Acronym: CARES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMX-67_301; U1111-1114-4194 (Registry Identifier: WHO)
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Results first posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular Outcomes; Heart Attack; Stroke; Drug Therapy; Physiology; Hyperuricemia; Uric Acid
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Stroke; Hyperuricemia | interventions — Febuxostat; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Febuxostat (Experimental): Febuxostat 40 mg (or 80 mg beginning on week 4 if serum uric acid level was ≥6.0 mg/dL), tablets, orally, once daily for up to approximately 82 months.
  Interventions: Drug: Febuxostat
- Allopurinol (Active Comparator): Allopurinol 300 mg to 600 mg (increased in 100 mg increments each month until serum uric acid was <6.0 mg/dL), tablets, orally, once daily for up to approximately 83 months to participants with mildly impaired renal function or normal renal function (estimated creatinine clearance [eCLcr] ≥60 mL/min) or allopurinol 200 mg to 400 mg (increased in 100 mg increments each month until serum uric acid was <6.0 mg/dL), tablets, orally, once daily for up to approximately 83 months to participants with moderately impaired renal function (eCLcr ≥30 but <60 mL/min).
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Febuxostat — Febuxostat tablets
  Other Names: Uloric; TMX-67
  Arms: Febuxostat
Drug: Allopurinol — Allopurinol tablets
  Other Names: Zyloprim; Allohexal; Allosig; Milurit; Alloril; Progout; Zyloric; Puricos; Zyrik 300; Aluron
  Arms: Allopurinol

SUMMARY:
The purpose of this study is to see whether subjects with gout who receive febuxostat or allopurinol for up to 9 years have a higher rate of serious heart and blood vessel complications (major cardiovascular events).

DETAILED DESCRIPTION:
The drug tested in this study was called Febuxostat (TMX-67). Febuxostat compared with allopurinol was evaluated for the cardiovascular (CV) safety in people with gout and significant CV comorbidities.

The study enrolled 6198 patients. Participants with a diagnosis of gout were enrolled in a 1:1 ratio to receive either:

* Febuxostat
* Allopurinol

Participants received febuxostat 40 mg or 80 mg for the study depending on their serum uric acid levels were either <6.0 mg/dL or ≥6.0 mg/dL during specified visits. Allopurinol 200 mg to 400 mg (for moderate renal impairment),or 300 mg to 600 mg (for normal and mild renal impairment), increased in 100 mg increments each month until serum uric acid was <6.0 mg/dL was received.

This multi-center trial was conducted in Canada, Mexico and United States. The overall time to participate in this study was approximately 7 years (84 months). Participants made multiple visits to the clinic and were also contacted through the telephone.

ELIGIBILITY:
Inclusion Criteria:

1. The participant or the participant's legally acceptable representative signs and dates a written, informed consent form/Health Insurance Portability and Accountability Act (HIPAA) Authorization prior to the initiation of any study procedures.
2. The participant is male ≥50 years of age or female ≥55 years of age and at least 2-years post-menopausal.
3. The participant has a history of major CV or cerebrovascular disease including at least one of the following:

   * Myocardial infarction (MI).
   * Hospitalized unstable angina.
   * Cardiac or cerebrovascular revascularization procedure.
   * Stroke.
   * Hospitalized transient ischemic attack (TIA).
   * Peripheral vascular disease (ankle brachial index ≤0.6, revascularization and/or well-documented history of claudication).
   * History of diabetes mellitus with evidence of micro- or macrovascular disease (retinopathy, neuropathy, nephropathy, small vessel vascular diseases).
4. The participant has a history or presence of gout defined as having one or more of the American Rheumatism Association criteria for the diagnosis of gout:

   * A tophus proven to contain urate crystals by chemical or polarized light microscopic means, and/or
   * Characteristic urate crystals in the joint fluid, and/or
   * History of at least 6 of the following clinical, laboratory, and X-ray phenomena:

     * More than 1 attack of acute arthritis.
     * Maximum inflammation developed within 1 day.
     * Monoarticular arthritis.
     * Redness observed over joints.
     * First metatarsophalangeal joint painful or swollen.
     * Unilateral first metatarsophalangeal joint attack.
     * Unilateral tarsal joint attack.
     * Tophus (proven or suspected).
     * Hyperuricemia.
     * Asymmetric swelling within a joint on x-ray.
     * Subcortical cysts without erosions on x-ray.
     * Joint fluid culture negative for organisms during attack.
5. The participants must have either:

   * a serum urate or serum uric acid (sUA) level ≥7.0 mg/dL (≥416 μmol/L) at the Day -7 Visit OR
   * a sUA level ≥6.0 mg/dL (≥354 μmol/L) at the Day -7 Visit AND inadequately controlled gout (≥1 flare in the 12 months prior to screening and/or the presence of tophi).
6. The participant is capable of understanding and complying with protocol requirements

Exclusion Criteria:

Participants who meet any of the following criteria will not qualify for entry into this study:

1. The participant has secondary hyperuricemia (eg, due to myeloproliferative disorder, or organ transplant).
2. The participant has a history of xanthinuria.
3. The participant has received urate-lowering therapy (i.e., febuxostat, allopurinol, probenecid, etc.) or excluded medication during the screening period (beginning with Day -7).
4. The participant has a known hypersensitivity to febuxostat or allopurinol or any components of their formulation.
5. The participant has active peptic ulcer disease.
6. The participant has a history of cancer (other than basal cell carcinoma of the skin) within 5 years prior to the first dose of study medication.
7. The participant had MI or stroke within 60 days prior to the Screening Visit.
8. The participant has alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) values greater than 2 times the upper limit of normal (×ULN) during the Screening period.
9. The participant has a significant medical condition and/or conditions that would interfere with the treatment, safety, or compliance with the protocol.
10. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 5 years prior to the Screening Visit or the participant consumes >14 alcoholic beverages per week.
11. The participant has received any investigational medicinal product within the 30 days prior to the Screening Visit and throughout the study.
12. The participant's estimated creatinine clearance (CLcr) is <30 mL/min, where CLcr is calculated using the Cockcroft and Gault formula based on ideal body weight (IBW),
13. The participant is an immediate family member, study site employee, or is in a dependant relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
14. The participant is required to take excluded medications
15. The participant has a known history of infection with hepatitis B, hepatitis C, or human immunodeficiency virus.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6198 (Actual)
Dates: Start 2010-04-23 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (203):
- United States (202):
  - Decatur, Georgia
  - Dunwoody, Georgia
  - Marietta, Georgia
  - Norcross, Georgia
  - Roswell, Georgia
  - Suwanee, Georgia
  - Waycross, Georgia
  - Honolulu, Hawaii
  - Boise, Idaho
  - Coeur d'Alene, Idaho
  - Nampa, Idaho
  - Addison, Illinois
  - Arlington Heights, Illinois
  - Evanston, Illinois
  - Evergreen Park, Illinois
  - Flossmoor, Illinois
  - Melrose Park, Illinois
  - Morton, Illinois
  - Naperville, Illinois
  - Quincy, Illinois
  - Rockford, Illinois
  - Bloomington, Indiana
  - Brownsburg, Indiana
  - Lafayette, Indiana
  - Valparaiso, Indiana
  - Iowa City, Iowa
  - Lenexa, Kansas
  - Overland Park, Kansas
  - Topeka, Kansas
  - Wichita, Kansas
  - Elizabethtown, Kentucky
  - Lexington, Kentucky
  - Owensboro, Kentucky
  - Paducah, Kentucky
  - Mer Rouge, Louisiana
  - Monroe, Louisiana
  - Shreveport, Louisiana
  - Biddeford, Maine
  - Rockport, Maine
  - Baltimore, Maryland
  - Cumberland, Maryland
  - Hagerstown, Maryland
  - Lutherville, Maryland
  - Wheaton, Maryland
  - Brockton, Massachusetts
  - Fall River, Massachusetts
  - Hyannis, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Bingham Farms, Michigan
  - Chelsea, Michigan
  - Detroit, Michigan
  - Flint, Michigan
  - Kalamazoo, Michigan
  - Lansing, Michigan
  - Chaska, Minnesota
  - Duluth, Minnesota
  - Edina, Minnesota
  - Saint Paul, Minnesota
  - Jackson, Mississippi
  - Olive Branch, Mississippi
  - Port Gibson, Mississippi
  - Clarkson Valley, Missouri
  - Hazelwood, Missouri
  - Kansas City, Missouri
  - Saint Charles, Missouri
  - St Louis, Missouri
  - Washington, Missouri
  - Billings, Montana
  - Butte, Montana
  - Bellevue, Nebraska
  - Grand Island, Nebraska
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Henderson, Nevada
  - Las Vegas, Nevada
  - Reno, Nevada
  - Brick, New Jersey
  - Edison, New Jersey
  - Oradell, New Jersey
  - Albuquerque, New Mexico
  - Las Vegas, New Mexico
  - Endwell, New York
  - Freeport, New York
  - Glens Falls, New York
  - Mineola, New York
  - New Windsor, New York
  - New York, New York
  - Rochester, New York
  - West Seneca, New York
  - Westfield, New York
  - Asheboro, North Carolina
  - Cary, North Carolina
  - Charlotte, North Carolina
  - Columbia, North Carolina
  - Greensboro, North Carolina
  - Huntersville, North Carolina
  - Lenoir, North Carolina
  - Monroe, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Shelby, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Akron, Ohio
  - Centerville, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Delaware, Ohio
  - Franklin, Ohio
  - Kettering, Ohio
  - Lyndhurst, Ohio
  - Marion, Ohio
  - Mentor, Ohio
  - Middleburg Heights, Ohio
  - Toledo, Ohio
  - Willoughby Hills, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Ashland, Oregon
  - Bend, Oregon
  - Eugene, Oregon
  - Portland, Oregon
  - Altoona, Pennsylvania
  - Bensalem, Pennsylvania
  - Bethlehem, Pennsylvania
  - Downingtown, Pennsylvania
  - Duncansville, Pennsylvania
  - Ephrata, Pennsylvania
  - Harleysville, Pennsylvania
  - Lansdale, Pennsylvania
  - McMurray, Pennsylvania
  - Philadelphia, Pennsylvania
  - Quakertown, Pennsylvania
  - Wyomissing, Pennsylvania
  - Cumberland, Rhode Island
  - East Providence, Rhode Island
  - Providence, Rhode Island
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Greenville, South Carolina
  - Greenwood, South Carolina
  - Greer, South Carolina
  - Myrtle Beach, South Carolina
  - Orangeburg, South Carolina
  - Pelzer, South Carolina
  - Simpsonville, South Carolina
  - Spartanburg, South Carolina
  - Athens, Tennessee
  - Chattanooga, Tennessee
  - Clarksville, Tennessee
  - Collierville, Tennessee
  - Fayetteville, Tennessee
  - Jackson, Tennessee
  - Kingsport, Tennessee
  - Memphis, Tennessee
  - New Tazewell, Tennessee
  - Bellaire, Texas
  - Carrollton, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Fort Worth, Texas
  - Grapevine, Texas
  - Houston, Texas
  - Irving, Texas
  - McKinney, Texas
  - New Braunfels, Texas
  - Odessa, Texas
  - Pearland, Texas
  - Plano, Texas
  - Richardson, Texas
  - San Antonio, Texas
  - Southlake, Texas
  - Sugar Land, Texas
  - Tomball, Texas
  - Waco, Texas
  - Bountiful, Utah
  - Draper, Utah
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Alexandria, Virginia
  - Arlington, Virginia
  - Burke, Virginia
  - Danville, Virginia
  - McLean, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Salem, Virginia
  - Virginia Beach, Virginia
  - Port Orchard, Washington
  - Tacoma, Washington
  - Clarksburg, West Virginia
  - Green Bay, Wisconsin
  - Milwaukee, Wisconsin
  - New Berlin, Wisconsin
  - Oregon, Wisconsin
  - Verona, Wisconsin
  - Waukesha, Wisconsin
  - Weston, Wisconsin
- Jalisco, Mexico City, Mexico

REFERENCES:
- [Result] White WB, Chohan S, Dabholkar A, Hunt B, Jackson R. Cardiovascular safety of febuxostat and allopurinol in patients with gout and cardiovascular comorbidities. Am Heart J. 2012 Jul;164(1):14-20. doi: 10.1016/j.ahj.2012.04.011. Epub 2012 Jun 13. PMID 22795277
- [Result] White WB, Saag KG, Becker MA, Borer JS, Gorelick PB, Whelton A, Hunt B, Castillo M, Gunawardhana L; CARES Investigators. Cardiovascular Safety of Febuxostat or Allopurinol in Patients with Gout. N Engl J Med. 2018 Mar 29;378(13):1200-1210. doi: 10.1056/NEJMoa1710895. Epub 2018 Mar 12. PMID 29527974
- [Derived] Saag KG, Becker MA, White WB, Whelton A, Borer JS, Gorelick PB, Hunt B, Castillo M, Gunawardhana L; CARES Investigators. Evaluation of the Relationship Between Serum Urate Levels, Clinical Manifestations of Gout, and Death From Cardiovascular Causes in Patients Receiving Febuxostat or Allopurinol in an Outcomes Trial. Arthritis Rheumatol. 2022 Sep;74(9):1593-1601. doi: 10.1002/art.42160. Epub 2022 Aug 5. PMID 35536764
- [Derived] Fravel MA, Ernst ME. Management of gout in the older adult. Am J Geriatr Pharmacother. 2011 Oct;9(5):271-85. doi: 10.1016/j.amjopharm.2011.07.004. Epub 2011 Aug 17. PMID 21849262
- See also: Uloric Package Insert — http://general.takedapharm.com/content/file.aspx?applicationcode=6C7C39D8-5D09-453B-BF30-696A4AB88E62&fileTypeCode=ULORICPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 320 investigative sites in Canada, Mexico and United States from 23 April 2010 to 18 July 2017.
Pre-assignment Details: Participants with a diagnosis of gout and significant cardiovascular comorbidities were enrolled in a 1:1 ratio to receive either febuxostat or allopurinol.
Period: Overall Study
Arm/Group | Febuxostat | Allopurinol
Started | 3101 | 3097
Completed | 1704 | 1706
Not Completed | 1397 | 1391
Not completed — Adverse Event | 191 | 172
Not completed — Major Protocol Deviation | 52 | 46
Not completed — Lost to Follow-up | 226 | 223
Not completed — Voluntary Withdrawal | 595 | 587
Not completed — Reason not Specified | 333 | 363

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who were randomized and received at least 1 dose of double-blind study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Febuxostat | Allopurinol | Total
Number analyzed (Participants) | 3098 | 3092 | 6190
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (8.58) | 65.0 (8.49) | 64.8 (8.53)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 1584 | 1506 | 3090
  65 to <75 years | 1094 | 1135 | 2229
  ≥75 years | 420 | 451 | 871
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 494 | 500 | 994
  Male | 2604 | 2592 | 5196
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 262 | 234 | 496
  Asian | 92 | 96 | 188
  Black or African American | 552 | 593 | 1145
  Native Hawaiian or Other Pacific Islander | 13 | 14 | 27
  White | 2160 | 2140 | 4300
  Other | 19 | 15 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 539 | 521 | 1060
  Not Hispanic or Latino | 2559 | 2571 | 5130
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 68 | 72 | 140
  Mexico | 379 | 355 | 734
  United States | 2651 | 2665 | 5316
Height [Mean (Standard Deviation); unit: cm] | 172.9 (9.54) | 173.0 (9.77) | 173.0 (9.65)
Weight [Mean (Standard Deviation); unit: kg] — Population: Here, number analyzed indicates participants who were evaluated for this baseline characteristic.
  kg
    number analyzed (Participants) | 3098 | 3087 | 6185
    (all) | 100.5 (22.47) | 100.3 (22.89) | 100.4 (22.68)
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2] Population: Here, number analyzed indicates participants who were evaluated for this baseline characteristic.
  kg/m^2
    number analyzed (Participants) | 3098 | 3087 | 6185
    (all) | 32.5 [18 to 73] | 32.1 [17 to 75] | 32.3 [17 to 75]
BMI Categorical [Count of Participants; unit: Participants] — Body Mass Index = weight (kg)/[height (m)^2]
  Participants
    <25 | 201 | 201 | 402
    25-30 | 844 | 862 | 1706
    ≥30 | 2053 | 2024 | 4077
Smoking History [Count of Participants; unit: Participants]
  Never smoked | 1175 | 1124 | 2299
  Ex-smoker | 1533 | 1553 | 3086
  Current smoker | 390 | 415 | 805
Alcohol History [Count of Participants; unit: Participants]
  Never drank | 792 | 784 | 1576
  Ex-drinker | 805 | 812 | 1617
  Current drinker | 1501 | 1496 | 2997
Renal Function [Count of Participants; unit: Participants] — Moderate renal impairment: eCLcr=30 to 59 mL/min; mild renal impairment: eCLcr=60 to 89 mL/min; normal: eCLcr ≥90 mL/min. Seven subjects with Baseline eCLcr <30 mL/min and 1 subject with missing Baseline eCLcr
  Participants
    Moderately Impaired | 1636 | 1631 | 3267
    Mildly Impaired | 1217 | 1231 | 2448
    Normal | 239 | 228 | 467
History of Kidney Stone [Count of Participants; unit: Participants]
  Yes | 627 | 627 | 1254
  No | 2471 | 2465 | 4936
Use of Low Dose Aspirin [Count of Participants; unit: Participants] — Dosing <325 mg aspirin per day is considered as low-dose aspirin
  Participants
    Yes | 1496 | 1481 | 2977
    No | 1602 | 1611 | 3213
Use of any Dose of Aspirin [Count of Participants; unit: Participants]
  Yes | 1894 | 1933 | 3827
  No | 1204 | 1159 | 2363
Use of Nonsteroidal Anti-Inflammatory Drug (NSAIDs) [Count of Participants; unit: Participants]
  Yes | 856 | 908 | 1764
  No | 2242 | 2184 | 4426
Use of Clopidogrel and Other Antiplatelet Drugs [Count of Participants; unit: Participants]
  Yes | 599 | 627 | 1226
  No | 2499 | 2465 | 4964

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Primary Major Adverse Cardiovascular Events (MACE) Composite (75% Interim Analysis)
Description: Major adverse cardiovascular events (MACE) were defined as a composite of cardiovascular (CV) death, non-fatal myocardial infarction (MI), nonfatal stroke and unstable angina with urgent coronary revascularization; these events were adjudicated by an independent cardiovascular endpoints committee.
Time Frame: Up to last dose of study drug (approximately 83 months)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Febuxostat | Allopurinol
Number analyzed (Participants) | 3039 | 3034
percentage of participants | 8.0 | 8.0
Statistical Analysis 1: Comparison: Febuxostat vs Allopurinol; Statistical analysis for the primary endpoint was based on 1-sided repeated confidence intervals (CIs), using critical values from a 1-sided stopping boundary for a group sequential design (GSD), to preserve an overall false-rejection rate of 2.5%, to assess non-inferiority at each interim analysis and the final analysis; Test type: Non-Inferiority — Noninferiority was declared if the upper 1-sided CI for the hazard ratio was less than 1.3. Critical boundary of 2.359 (75% interim) based on the Lan-DeMets-O'Brien-Fleming alpha spending function was used for CI estimation; Cox Proportional Hazard = 0.99, 97% CI 1-sided [upper limit 1.23] — Time from randomization to the first occurrence of any MACE was fitted using Cox Proportional Hazard model with treatment as a covariate and Baseline renal function as a stratification factor

2. Secondary Outcome: Percentage of Participants With Antiplatelet Trialists' Collaborative (APTC) Event
Description: APTC events were defined as a composite of cardiovascular death, nonfatal myocardial infarction, and nonfatal stroke; these events were adjudicated by an independent cardiovascular endpoints committee.
Time Frame: Up to last dose of study drug (approximately 83 months)
Population: FAS included all participants who were randomized and received at least 1 dose of double-blind study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Febuxostat | Allopurinol
Number analyzed (Participants) | 3098 | 3092
percentage of participants | 9.6 | 8.8
Statistical Analysis 1: Comparison: Febuxostat vs Allopurinol; Test type: Other; Cox Proportional Hazard = 1.09, 95% CI 2-sided [0.92 to 1.28] — Time from randomization to the first occurrence of any APTC event was fitted using Cox Proportional Hazard model with treatment as a covariate and Baseline renal function status as a stratification factor

3. Secondary Outcome: Percentage of Participants With Cardiovascular (CV) Death
Description: Events were adjudicated by an independent cardiovascular endpoints committee as CV death.
Time Frame: Up to last dose of study drug (approximately 83 months)
Population: FAS included all participants who were randomized and received at least 1 dose of double-blind study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Febuxostat | Allopurinol
Number analyzed (Participants) | 3098 | 3092
percentage of participants | 4.3 | 3.2
Statistical Analysis 1: Comparison: Febuxostat vs Allopurinol; Test type: Other; Cox Proportional Hazard = 1.34, 95% CI 2-sided [1.03 to 1.73] — Time from randomization to the first occurrence of cardiovascular death was fitted using Cox Proportional Hazard model with factors including treatment and baseline renal function

4. Secondary Outcome: Percentage of Participants With Non-fatal Myocardial Infarction (MI)
Description: Events were adjudicated by an independent cardiovascular endpoints committee as non-fatal MI.
Time Frame: Up to last dose of study drug (approximately 83 months)
Population: FAS included all participants who were randomized and received at least 1 dose of double-blind study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Febuxostat | Allopurinol
Number analyzed (Participants) | 3098 | 3092
percentage of participants | 3.6 | 3.8
Statistical Analysis 1: Comparison: Febuxostat vs Allopurinol; Test type: Other; Cox Proportional Hazard = 0.93, 95% CI 2-sided [0.72 to 1.21] — Time from randomization to the first occurrence of non-fatal MI was fitted using Cox Proportional Hazard model with factors including treatment and baseline renal function

5. Secondary Outcome: Percentage of Participants With Non-fatal Stroke
Description: Events were adjudicated by an independent cardiovascular endpoints committee as non-fatal stroke.
Time Frame: Up to last dose of study drug (approximately 83 months)
Population: FAS included all participants who were randomized and received at least 1 dose of double-blind study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Febuxostat | Allopurinol
Number analyzed (Participants) | 3098 | 3092
percentage of participants | 2.3 | 2.3
Statistical Analysis 1: Comparison: Febuxostat vs Allopurinol; Test type: Other; Cox Proportional Hazard = 1.01, 95% CI 2-sided [0.73 to 1.41] — Time from randomization to the first occurrence of non-fatal stroke was fitted using Cox Proportional Hazard model with factors including treatment and baseline renal function

6. Secondary Outcome: Percentage of Participants With Unstable Angina With Urgent Coronary Revascularization
Description: Events were adjudicated by an independent cardiovascular endpoints committee as unstable angina with urgent coronary revascularization.
Time Frame: Up to last dose of study drug (approximately 83 months)
Population: FAS included all participants who were randomized and received at least 1 dose of double-blind study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Febuxostat | Allopurinol
Number analyzed (Participants) | 3098 | 3092
percentage of participants | 1.6 | 1.8
Statistical Analysis 1: Comparison: Febuxostat vs Allopurinol; Test type: Other; Cox Proportional Hazard = 0.86, 95% CI 2-sided [0.59 to 1.26] — Time from randomization to the first occurrence of unstable angina with urgent coronary revascularization was fitted using Cox Proportional Hazard model with factors including treatment and baseline renal function

7. Primary Outcome: Percentage of Participants With Primary MACE Composite (Final Analysis)
Description: as for outcome 1
Time Frame: Up to last dose of study drug (approximately 83 months)
Population: FAS included all participants who were randomized and received at least 1 dose of double-blind study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Febuxostat | Allopurinol
Number analyzed (Participants) | 3098 | 3092
percentage of participants | 10.8 | 10.4
Statistical Analysis 1: Comparison: Febuxostat vs Allopurinol; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — Noninferiority was declared if the upper 1-sided CI for the hazard ratio was less than 1.3. Critical boundary of 2.014 (final analysis) based on the Lan-DeMets-O'Brien-Fleming alpha spending function was used for CI estimation; Cox Proportional Hazard = 1.03, 97% CI 2-sided [0.87 to 1.23] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: First dose of study drug to 30 days after last dose of study drug (Approximately 84 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Febuxostat | Allopurinol
All-Cause Mortality (participants affected / at risk) | 243/3098 | 199/3092
Serious Adverse Events (participants affected / at risk) | 1046/3098 | 995/3092
Other Adverse Events (participants affected / at risk) | 1450/3098 | 1467/3092
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Febuxostat (N=3098) | Allopurinol (N=3092)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 17 | 15
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 3 | 3
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 3 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Aortic valve calcification (Cardiac disorders) | 0 | 1
Aortic valve disease (Cardiac disorders) | 1 | 1
Aortic valve incompetence (Cardiac disorders) | 2 | 2
Aortic valve sclerosis (Cardiac disorders) | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 4
Atrioventricular block complete (Cardiac disorders) | 4 | 5
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 2 | 1
Bifascicular block (Cardiac disorders) | 1 | 0
Defect conduction intraventricular (Cardiac disorders) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 0 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 3 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Cardiovascular disorder (Cardiac disorders) | 1 | 1 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 3 | 1 — Three treatment-emergent deaths occurred during treatment with febuxostat and are not related.
Malignant hypertensive heart disease (Cardiac disorders) | 0 | 1
Cardiac discomfort (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1
Cardiac valve disease (Cardiac disorders) | 0 | 1
Heart valve incompetence (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 4 | 3
Congestive cardiomyopathy (Cardiac disorders) | 2 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 12 | 7 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Arteriosclerosis coronary artery (Cardiac disorders) | 4 | 4 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Coronary artery disease (Cardiac disorders) | 51 | 58 — Two treatment-emergent deaths occurred during treatment with febuxostat and are not related; Two treatment-emergent deaths occurred during treatment with allopurinol and are not related.
Coronary artery occlusion (Cardiac disorders) | 7 | 8
Coronary artery stenosis (Cardiac disorders) | 2 | 7
Cardiac failure (Cardiac disorders) | 8 | 9 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Cardiac failure acute (Cardiac disorders) | 8 | 9 — Two treatment-emergent deaths occurred during treatment with febuxostat and are not related.
Cardiac failure chronic (Cardiac disorders) | 4 | 5 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Cardiac failure congestive (Cardiac disorders) | 124 | 109 — Ten treatment-emergent deaths occurred during treatment with febuxostat and are not related; Eight treatment-emergent deaths occurred during treatment with allopurinol and are not related.
Cardiogenic shock (Cardiac disorders) | 5 | 5 — Two treatment-emergent deaths occurred during treatment with febuxostat and are not related; One treatment-emergent death occurred during treatment with allopurinol and is not related.
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Ventricular failure (Cardiac disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 6 | 8 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Acute myocardial infarction (Cardiac disorders) | 63 | 68 — Five treatment-emergent deaths occurred during treatment with febuxostat and are not related; Two treatment-emergent deaths occurred during treatment with allopurinol and are not related.
Angina unstable (Cardiac disorders) | 34 | 33
Myocardial infarction (Cardiac disorders) | 41 | 51 — Eleven treatment-emergent deaths occurred during treatment with febuxostat and are not related; Seven treatment-emergent deaths occurred during treatment with allopurinol and are not related.
Myocardial ischaemia (Cardiac disorders) | 8 | 5 — One treatment-emergent death occurred during treatment with febuxostat and is not related; Two treatment-emergent deaths occurred during treatment with allopurinol and are not related.
Silent myocardial infarction (Cardiac disorders) | 2 | 0
Subendocardial ischaemia (Cardiac disorders) | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 6 | 0
Mitral valve prolapse (Cardiac disorders) | 2 | 0
Cardiac aneurysm (Cardiac disorders) | 0 | 1
Cardiac hypertrophy (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 2 | 1
Systolic dysfunction (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 4 | 6 — Two treatment-emergent deaths occurred during treatment with febuxostat and are not related.
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 12 | 6
Chronotropic incompetence (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 8 | 5
Cor pulmonale (Cardiac disorders) | 0 | 2 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Right ventricular failure (Cardiac disorders) | 1 | 2 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 65 | 64 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Atrial flutter (Cardiac disorders) | 10 | 12 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Atrial tachycardia (Cardiac disorders) | 1 | 1
Sinus bradycardia (Cardiac disorders) | 2 | 2
Sinus node dysfunction (Cardiac disorders) | 8 | 6
Sinus tachycardia (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 5 | 4
Accelerated idioventricular rhythm (Cardiac disorders) | 0 | 2
Cardiac arrest (Cardiac disorders) | 17 | 11 — Eleven treatment-emergent deaths occurred during treatment with febuxostat and are not related; Eight treatment-emergent deaths occurred during treatment with allopurinol and are not related.
Cardio-respiratory arrest (Cardiac disorders) | 4 | 2 — Four treatment-emergent deaths occurred during treatment with febuxostat and are not related; Two treatment-emergent deaths occurred during treatment with allopurinol and are not related.
Pulseless electrical activity (Cardiac disorders) | 1 | 1 — One treatment-emergent death occurred during treatment with febuxostat and is not related; One treatment-emergent death occurred during treatment with allopurinol and is not related.
Ventricular arrhythmia (Cardiac disorders) | 1 | 3 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 4 | 6 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Ventricular tachyarrhythmia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 25 | 25 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Cystic lymphangioma (Congenital, familial and genetic disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 4 | 3
Vertigo positional (Ear and labyrinth disorders) | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Thyroid mass (Endocrine disorders) | 1 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Blindness unilateral (Eye disorders) | 1 | 0
Sudden visual loss (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 2
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 7 | 3
Pancreatitis acute (Gastrointestinal disorders) | 4 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0
Duodenal polyp (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 3 | 2
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0
Poor dental condition (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 4
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 3
Small intestinal obstruction (Gastrointestinal disorders) | 9 | 5
Volvulus of small bowel (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 3 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 2 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 8 | 11
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 2
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 6
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 1 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 4 | 4
Oesophageal food impaction (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 4 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Intussusception (Gastrointestinal disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 1
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 2 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 2
Colonic haematoma (Gastrointestinal disorders) | 1 | 0
Mesenteric haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 4
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 2 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Rectal adenocarcinoma (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 0 | 2
Vomiting projectile (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 18 | 17 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Haematemesis (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 4
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 3
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 2 | 4
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 2 | 1
Asthenia (General disorders) | 4 | 8
Fatigue (General disorders) | 2 | 0
Medical device pain (General disorders) | 0 | 2
Accidental death (General disorders) | 0 | 1 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Death (General disorders) | 5 | 1 — Five treatment-emergent deaths occurred during treatment with febuxostat and are not related; One treatment-emergent death occurred during treatment with allopurinol and is not related.
Drowning (General disorders) | 1 | 0 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Sudden cardiac death (General disorders) | 1 | 2 — One treatment-emergent death occurred during treatment with febuxostat and is not related; Two treatment-emergent deaths occurred during treatment with allopurinol and are not related.
Sudden death (General disorders) | 1 | 0 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Pyrexia (General disorders) | 3 | 3
Condition aggravated (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Local swelling (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Impaired healing (General disorders) | 2 | 0
Strangulated hernia (General disorders) | 0 | 1
Implant site inflammation (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 3 | 0 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Haemorrhagic cyst (General disorders) | 1 | 0
Necrobiosis (General disorders) | 0 | 1
Generalised oedema (General disorders) | 3 | 2
Oedema (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 2 | 1
Chest discomfort (General disorders) | 4 | 8
Chest pain (General disorders) | 25 | 25
Non-cardiac chest pain (General disorders) | 34 | 32
Pain (General disorders) | 0 | 1
Surgical failure (General disorders) | 1 | 3
Ulcer haemorrhage (General disorders) | 0 | 1
Vascular stent occlusion (General disorders) | 0 | 1
Vascular stent restenosis (General disorders) | 1 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 6 | 7
Cholecystitis acute (Hepatobiliary disorders) | 7 | 8
Cholecystitis chronic (Hepatobiliary disorders) | 2 | 1
Cholelithiasis (Hepatobiliary disorders) | 5 | 9
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 2 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 4
Hepatic haematoma (Hepatobiliary disorders) | 1 | 0
Granulomatous liver disease (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 2 | 2
Sarcoidosis (Immune system disorders) | 1 | 1
Drug hypersensitivity (Immune system disorders) | 2 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 1
Abdominal abscess (Infections and infestations) | 0 | 2
Abdominal wall abscess (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 3 | 1
Appendicitis perforated (Infections and infestations) | 0 | 1
Colonic abscess (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 7 | 9
Gastroenteritis (Infections and infestations) | 7 | 7
Perirectal abscess (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 2
Bacterial infection (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 3 | 0
Bronchitis bacterial (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 30 | 21
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 4 | 2
Gastroenteritis bacterial (Infections and infestations) | 0 | 1
Incisional hernia gangrenous (Infections and infestations) | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 1
Oral bacterial infection (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 3 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Arthritis infective (Infections and infestations) | 0 | 1
Bursitis infective (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 15 | 9 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Osteomyelitis acute (Infections and infestations) | 0 | 1
Pertussis (Infections and infestations) | 1 | 0
Lyme disease (Infections and infestations) | 0 | 1
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 2
CNS ventriculitis (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 3 | 2
Clostridium difficile infection (Infections and infestations) | 2 | 3
Gas gangrene (Infections and infestations) | 1 | 0
Sialoadenitis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Labyrinthitis (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 2 | 0
Vulval abscess (Infections and infestations) | 0 | 1
Helicobacter gastritis (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 1
Herpes simplex meningitis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 2 | 0
Herpes zoster meningomyelitis (Infections and infestations) | 1 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 2
Abscess rupture (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 2 | 1
Empyema (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 0 | 1
Groin infection (Infections and infestations) | 1 | 1
Implant site infection (Infections and infestations) | 0 | 2
Incision site infection (Infections and infestations) | 1 | 0
Infected bite (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 2
Injection site infection (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 3 | 3
Mediastinitis (Infections and infestations) | 1 | 1
Medical device site infection (Infections and infestations) | 1 | 0
Postoperative abscess (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 3 | 0
Wound infection (Infections and infestations) | 2 | 3
Influenza (Infections and infestations) | 9 | 3 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Pneumonia legionella (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 10 | 9
Infectious pleural effusion (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 67 | 88 — One treatment-emergent death occurred during treatment with febuxostat and is not related; Six treatment-emergent deaths occurred during treatment with allopurinol and are not related.
Pneumonia necrotising (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Proteus infection (Infections and infestations) | 2 | 0
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 6 | 4
Device related sepsis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 24 | 24 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Septic embolus (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 7 | 10 — Two treatment-emergent deaths occurred during treatment with febuxostat and are not related; One treatment-emergent death occurred during treatment with allopurinol and is not related.
Urosepsis (Infections and infestations) | 9 | 4
Carbuncle (Infections and infestations) | 1 | 0
Diabetic foot infection (Infections and infestations) | 4 | 2
Infected skin ulcer (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 1 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 1
Endocarditis staphylococcal (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 3
Staphylococcal abscess (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 3
Staphylococcal infection (Infections and infestations) | 7 | 3
Staphylococcal parotitis (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 2 | 0
Beta haemolytic streptococcal infection (Infections and infestations) | 1 | 0
Cellulitis streptococcal (Infections and infestations) | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 2 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 2 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Cellulitis pharyngeal (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Cystitis (Infections and infestations) | 0 | 2
Kidney infection (Infections and infestations) | 2 | 2
Pyelonephritis (Infections and infestations) | 0 | 4
Pyelonephritis acute (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 14 | 21
Lymphangitis (Infections and infestations) | 1 | 1
Bronchitis viral (Infections and infestations) | 0 | 1
Encephalitis viral (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 2 | 1
Pneumonia viral (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 3
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 | 0 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Vascular injury (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 2 | 0
Epidural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 4
Subdural haematoma (Injury, poisoning and procedural complications) | 4 | 6 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 | 0
Open globe injury (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 3
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Open fracture (Injury, poisoning and procedural complications) | 0 | 1
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 2 | 2
Foot fracture (Injury, poisoning and procedural complications) | 2 | 1
Hand fracture (Injury, poisoning and procedural complications) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 6 | 6 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 2
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 2
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 3
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 2 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 0
Psychosis postoperative (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 7 | 13 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 5 | 5 — Three treatment-emergent deaths occurred during treatment with febuxostat and are not related; One treatment-emergent death occurred during treatment with allopurinol and is not related.
Wound (Injury, poisoning and procedural complications) | 0 | 2
Failure to anastomose (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 2 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 3
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 4 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1 | 0
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 5 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Scrotal haematoma (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 2 | 2
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 3
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 3 | 4
Blood glucose decreased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 1
Ejection fraction decreased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Prothrombin time ratio decreased (Investigations) | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1
Occult blood positive (Investigations) | 0 | 1
Heart rate increased (Investigations) | 1 | 0
Heart rate irregular (Investigations) | 2 | 0
Computerised tomogram abnormal (Investigations) | 0 | 1
Laboratory test abnormal (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 2
Liver function test increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 1
Blood creatine increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 1
Cardioactive drug level increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 1
Influenza B virus test positive (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 5 | 3
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2
Diabetic complication (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 2 | 1
Gout (Metabolism and nutrition disorders) | 4 | 6
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Hyperosmolar state (Metabolism and nutrition disorders) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 3 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 12 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 9 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 3
Dehydration (Metabolism and nutrition disorders) | 22 | 23
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 3 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Arthritis (Musculoskeletal and connective tissue disorders) | 12 | 7
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 3 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 | 3
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 2
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 5
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 4
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 7
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 5 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 40 | 34
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 5 | 3
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 6 | 6
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 6 | 3
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 2
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 3 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleomorphic malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 — One treatment-emergent death occurred during treatment with febuxostat and is not related; One treatment-emergent death occurred during treatment with allopurinol and is not related.
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 — One treatment-emergent death occurred during treatment with febuxostat and is not related; One treatment-emergent death occurred during treatment with allopurinol and is not related.
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 — One treatment-emergent death occurred during treatment with febuxostat and is not related; One treatment-emergent death occurred during treatment with allopurinol and is not related.
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Adenosquamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Lung squamous cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant neoplasm of eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 — Three treatment-emergent deaths occurred during treatment with febuxostat and are not related; One treatment-emergent death occurred during treatment with allopurinol and is not related.
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 — One treatment-emergent death occurred during treatment with febuxostat and is not related; Two treatment-emergent deaths occurred during treatment with allopurinol and are not related.
Squamous cell carcinoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Kidney angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 — One treatment-emergent death occurred during treatment with febuxostat and is not related; Two treatment-emergent deaths occurred during treatment with allopurinol and are not related.
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 — Two treatment-emergent deaths occurred during treatment with febuxostat and are not related.
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5 — One treatment-emergent death occurred during treatment with febuxostat and is not related; Three treatment-emergent deaths occurred during treatment with allopurinol and are not related.
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Malignant melanoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Poorly differentiated thyroid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Petit mal epilepsy (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 3
Brain stem infarction (Nervous system disorders) | 1 | 0
Brain stem stroke (Nervous system disorders) | 2 | 0
Carotid artery occlusion (Nervous system disorders) | 1 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 1
Cerebral haematoma (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Cerebral infarction (Nervous system disorders) | 6 | 1 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 45 | 44 — One treatment-emergent death occurred during treatment with febuxostat and is not related; Two treatment-emergent deaths occurred during treatment with allopurinol and are not related.
Embolic stroke (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 2 | 6 — One treatment-emergent death occurred during treatment with febuxostat and is not related; Two treatment-emergent deaths occurred during treatment with allopurinol and are not related.
Haemorrhagic stroke (Nervous system disorders) | 2 | 1
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 3 | 3
Lacunar infarction (Nervous system disorders) | 1 | 3
Lacunar stroke (Nervous system disorders) | 0 | 1
Thalamic infarction (Nervous system disorders) | 0 | 1
Thalamus haemorrhage (Nervous system disorders) | 0 | 1
Thrombotic stroke (Nervous system disorders) | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 1
Carotid artery disease (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 7 | 10
Cervical myelopathy (Nervous system disorders) | 2 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 0 | 1
Diabetic coma (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 1
Dementia (Nervous system disorders) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 30 | 34
Loss of consciousness (Nervous system disorders) | 1 | 3
Encephalitis autoimmune (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 5 | 5
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Hepatic encephalopathy (Nervous system disorders) | 3 | 1
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 6
Toxic encephalopathy (Nervous system disorders) | 1 | 0
Uraemic encephalopathy (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Cluster headache (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 0 | 3
Hydrocephalus (Nervous system disorders) | 3 | 2
Normal pressure hydrocephalus (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 1
Sciatica (Nervous system disorders) | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 6 | 4
Presyncope (Nervous system disorders) | 10 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 2 | 2
Hemiparesis (Nervous system disorders) | 0 | 2
Paralysis (Nervous system disorders) | 0 | 1
Quadriparesis (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 7 | 11
Slow speech (Nervous system disorders) | 1 | 0
Nerve root compression (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 2 | 0
Spinal claudication (Nervous system disorders) | 0 | 1
Spinal cord disorder (Nervous system disorders) | 1 | 1
Spondylitic myelopathy (Nervous system disorders) | 0 | 1
Brain injury (Nervous system disorders) | 0 | 2
Cerebral ventricle dilatation (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 25 | 22
Device dislocation (Product Issues) | 1 | 0
Device failure (Product Issues) | 4 | 2
Device lead issue (Product Issues) | 0 | 1
Device battery issue (Product Issues) | 1 | 0
Device malfunction (Product Issues) | 0 | 1
Device occlusion (Product Issues) | 1 | 0
Device lead damage (Product Issues) | 0 | 1
Anxiety (Psychiatric disorders) | 3 | 3
Confusional state (Psychiatric disorders) | 2 | 5
Disorientation (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 2 | 0
Delirium tremens (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 1
Major depression (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 7 | 10
Panic attack (Psychiatric disorders) | 0 | 2
Shared psychotic disorder (Psychiatric disorders) | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 2 | 0
Substance use disorder (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 2 — Two treatment-emergent deaths occurred during treatment with allopurinol and are not related.
Intentional self-injury (Psychiatric disorders) | 0 | 2 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Suicidal behaviour (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 4 | 2
Bladder outlet obstruction (Renal and urinary disorders) | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 2
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0
Nephropathy (Renal and urinary disorders) | 0 | 1
Renal haematoma (Renal and urinary disorders) | 0 | 1
Renal mass (Renal and urinary disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 139 | 132 — Three treatment-emergent deaths occurred during treatment with allopurinol and are not related.
Chronic kidney disease (Renal and urinary disorders) | 8 | 4
End stage renal disease (Renal and urinary disorders) | 5 | 2
Renal failure (Renal and urinary disorders) | 19 | 19 — One treatment-emergent death occurred during treatment with febuxostat and is not related; One treatment-emergent death occurred during treatment with allopurinol and is not related.
Renal impairment (Renal and urinary disorders) | 7 | 3
Renal injury (Renal and urinary disorders) | 1 | 1
Malignant renal hypertension (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 8
Hydronephrosis (Renal and urinary disorders) | 3 | 2
Renal artery stenosis (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 2 | 5
Renal vein thrombosis (Renal and urinary disorders) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 2
Calculus bladder (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 2 | 4
Polyuria (Renal and urinary disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 2
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Pelvic haematoma (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 6 | 6
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 21
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 | 0 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 27 | 35
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 10
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Laryngeal dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 | 5 — One treatment-emergent death occurred during treatment with febuxostat and is not related; One treatment-emergent death occurred during treatment with allopurinol and is not related.
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 4 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 13 | 23 — One treatment-emergent death occurred during treatment with allopurinol and is not related.
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 4 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 5 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 20 | 14 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 34 | 43 — Seven treatment-emergent deaths occurred during treatment with febuxostat and are not related; One treatment-emergent death occurred during treatment with allopurinol and is not related.
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1 — One treatment-emergent death occurred during treatment with febuxostat and is not related. One treatment-emergent death occurred during treatment with allopurinol and is not related.
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 17 | 22 — Five treatment-emergent deaths occurred during treatment with febuxostat and are not related; Seven treatment-emergent death occurred during treatment with allopurinol and is not related.
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Blood blister (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Diabetic foot (Skin and subcutaneous tissue disorders) | 5 | 5
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 5
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Leg amputation (Surgical and medical procedures) | 0 | 1
Accelerated hypertension (Vascular disorders) | 3 | 0
Hypertensive crisis (Vascular disorders) | 10 | 3
Hypertensive emergency (Vascular disorders) | 2 | 1
Malignant hypertension (Vascular disorders) | 6 | 1
Aortic aneurysm (Vascular disorders) | 4 | 11
Aortic occlusion (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 9 | 3 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Leriche syndrome (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 2 | 0 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Shock (Vascular disorders) | 1 | 1 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Haematoma (Vascular disorders) | 6 | 3
Haemorrhage (Vascular disorders) | 2 | 0
Lymphoedema (Vascular disorders) | 0 | 2
Arterial thrombosis (Vascular disorders) | 0 | 1
Embolism venous (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 2
Arteriosclerosis (Vascular disorders) | 4 | 3 — One treatment-emergent death occurred during treatment with febuxostat and is not related; One treatment-emergent death occurred during treatment with allopurinol and is not related.
Peripheral venous disease (Vascular disorders) | 1 | 1
Vascular occlusion (Vascular disorders) | 0 | 1
Arterial rupture (Vascular disorders) | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 16 | 15
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 1 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 10 | 6
Dry gangrene (Vascular disorders) | 1 | 0
Iliac artery occlusion (Vascular disorders) | 2 | 0
Intermittent claudication (Vascular disorders) | 6 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 6 | 3
Peripheral artery occlusion (Vascular disorders) | 1 | 4
Peripheral artery stenosis (Vascular disorders) | 2 | 2
Peripheral ischaemia (Vascular disorders) | 7 | 1
Poor peripheral circulation (Vascular disorders) | 0 | 1
Aortic calcification (Vascular disorders) | 1 | 0
Essential hypertension (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 11 | 9
Hypotension (Vascular disorders) | 15 | 12
Arteriovenous fistula (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 5 | 7
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 16
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Angina pectoris (Cardiac disorders) | 74 | 59
Gastrointestinal angiodysplasia haemorrhagic (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Febuxostat (N=3098) | Allopurinol (N=3092)
Constipation (Gastrointestinal disorders) | 157 | 125
Diarrhoea (Gastrointestinal disorders) | 299 | 284
Nausea (Gastrointestinal disorders) | 156 | 132
Oedema peripheral (General disorders) | 168 | 183
Bronchitis (Infections and infestations) | 214 | 212
Upper respiratory tract infection (Infections and infestations) | 242 | 267
Urinary tract infection (Infections and infestations) | 146 | 180
Blood creatine phosphokinase increased (Investigations) | 148 | 161
Arthralgia (Musculoskeletal and connective tissue disorders) | 258 | 311
Back pain (Musculoskeletal and connective tissue disorders) | 216 | 187
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 137 | 159
Pain in extremity (Musculoskeletal and connective tissue disorders) | 222 | 218
Hypertension (Vascular disorders) | 209 | 261

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2013-08-27): https://cdn.clinicaltrials.gov/large-docs/35/NCT01101035/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT01101035/SAP_001.pdf